CLINICAL TRIAL: NCT04490200
Title: Effectiveness of a Novel Respirator With Chitosan Nanoparticles to Reduce the Incidence of SARS-CoV-2 Infection in Healthcare Professionals: Randomized Controlled Trial (VESTA Trial)
Brief Title: Effectiveness of a Novel Respirator With Chitosan Nanoparticles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brasilia (Other)
Collaborators: University of Campinas, Brazil (Other); Centro de Pesquisa em Biotecnologia Ltda (Industry); Hospital Regional da Asa Norte (HRAN) (Unknown)
Responsible Party: Principal Investigator, Prof. Rodrigo Luiz Carregaro, Principal Investigator, University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VESTA Trial; 32862320.0.0000.0030 (Other: Ethics Commitee FCE/UnB/CONEP)
Record Dates: First submitted 2020-07-19; First posted 2020-07-29 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Covid19; SARS-CoV Infection; Worker-Patient Transmission, Healthcare
Keywords: Protective personal equipment; SARS-Cov-2; Chitosan; Occupational health; Prevention
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled clinical trial, characterized by the application of semi facial respirators, in which participants will be randomly and concealed allocated into two groups: VESTA respirator (GExp) and Conventional N95 respirator (CG). The participants will be healthcare professionals working in hospital environments contaminated by SARS-Cov-2. The study will be reported following the recommendations of the CONSORT Statement.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The outcome assessor won't have any knowledge about the study purposes and will be unaware of the group allocation.
  Participants will be blinded as they will not distinguish the novel respirator (VESTA) from the conventional N95 respirator (both will have the same shape, color and size).
  The statistical analysis will also be performed blinded for group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novel chitosan semi facial respirator (VESTA) (Experimental): VESTA is a semi facial respirator that follows the same technical specifications of a N95 class PFF2 respirator. However, the VESTA respirator has nanoparticles in the filtering element, which is manufactured with a product of 50 gsm melt blown polypropylene-treated with an electrostatic charge. This filtering element deposits nanoparticles of polymeric biodegradable material known as chitosan. Chitosan can act as a surface for adsorption and viral inactivation.
  Interventions: Device: VESTA respirator
- Conventional N95 semi facial respirator (Active Comparator): The N95 PFF2 respirators are manufactured from TNT as defined in ABNT NBR 15052: 2004 and in the resolution of ANVISA RDC No. 356. The filtering element is usually formed by a layer of thin polypropylene fibers arranged at random. This configuration influences the particles (which constitute aerosols) to move along an extensive and tortuous path in relation to their size; thus, increasing the probability of them coming into contact with the fibers and being retained. A number of mechanisms influence the interception of particles by the fibers of the filter element. In addition to the mechanical interception mechanisms, the presence of charges on the surface of the filter material can enhance the association of particles with its fibers and optimize the efficiency of the respirator.
  Interventions: Device: Conventional N95 respirator

INTERVENTIONS:
Device: VESTA respirator — The protocol will be composed by the use of the VESTA respirator for 21 days (approximately 8 consecutive shifts lasting 6 to 12 hours, followed by approximately 36 hours of rest). Each participant will receive a total of approximately 8 respirators, with instructions for a maximum usage time of 6 hours. Therefore, participants will receive 1 respirator to be used in each shift of 6 hours, and 2 respirators in shifts of 12 hours. All participants will receive a booklet with guidelines and training in the use and proper handling of the respirator. All respirators will be sterilized and packaged in the laboratory, to ensure that they are not contaminated before use by the participants. The intervention will not change the participants' routine, considering that they already follow instructions for the use of protective personal equipment (PPE) and the proposed intervention will follow all local regulations and guidelines for the use and conservation of PPE and semi facial respirators.
  Arms: Novel chitosan semi facial respirator (VESTA)
Device: Conventional N95 respirator — The protocol will be composed by the use of the N95 respirator for 21 days (approximately 8 consecutive shifts lasting 6 to 12 hours, followed by approximately 36 hours of rest). Each participant will receive a total of approximately 8 respirators, with instructions for a maximum usage time of 6 hours. Therefore, participants will receive 1 respirator to be used in each shift of 6 hours, and 2 respirators in shifts of 12 hours. All participants will receive a booklet with guidelines and training in the use and proper handling of the respirator. All respirators will be sterilized and packaged in the laboratory, to ensure that they are not contaminated before use by the participants. The intervention will not change the participants' routine, considering that they already follow instructions for the use of protective personal equipment (PPE) and the proposed intervention will follow all local regulations and guidelines for the use and conservation of PPE and semi facial respirators.
  Arms: Conventional N95 semi facial respirator

SUMMARY:
The use of nanomaterials in semi-facial respirators could decrease the permeability of particles and promote a biocidal effect compared to conventional respirators (N95) and, therefore, to enhance the filtering power, aiming to mitigate harmful effects of bacteria and viruses. Chitosan is a natural cationic polymer derived from chitin, with characteristics such as being biodegradable, biocompatible, non-toxic, and presenting antimicrobial activity. This polymer has virucidal activity in several types of viruses, including other coronaviruses, given the attractive factor of its cationic charge for negative charges. The effectiveness of a novel individual protection semi-facial respirator (called VESTA) will be investigated, compared to a conventional N95 respirator. The respirators will be tested in healthcare professionals working in hospital environments and the effectiveness will be attributed to the lower incidence rate of infection by the SARS-CoV-2, and to the ability to filter these viruses after use by healthcare professionals exposed to potentially contaminated environments. The study will be carried out in two stages: i) Randomized Controlled Trial with reduced sample to confirm the sample size calculation (pilot trial), and ii) Randomized Controlled Trial (RCT). The RCT will be conducted with healthcare professionals who have contact with environments/patients infected by SARS-CoV-2 in hospital sectors with greater vulnerability to infection (urgency, emergency and intensive care units). The RCT will be conducted initially with a group of sixty participants (n = 30 in each group) for initial investigation of the potential for efficacy with the use of the respirators (VESTA and conventional N95) in two sectors (emergency and ICU) in a reference Hospital for COVID-19. The RCT will consist of two parallel groups: (1) Experimental Group (GExp) that will use the novel respirator (VESTA) and (2) Control Group (CG) that will use the standard respirator (N95). Participants will be recruited from participating hospitals and will be accompanied by 21 days in approximately eight consecutive shifts (ranging from shifts lasting 6 to 12 hours each, followed by approximately 36 hours of rest). Participants will be assessed at baseline (T0), at the end of the 10th day (T1), and at the end of the 21st day (T2).

DETAILED DESCRIPTION:
Context for the latest register update (May, 2022): Our randomized controlled pilot trial was conducted from February until April 2021, following the same methodological procedures described within the clinical trial register. After analyzing the data from the pilot trial we included some updates within the clinical trial register. Summary of changes after the pilot trial: 1) We performed a new sample size calculation, which resulted in a sample size of 700 participants (n=350 in each group). This information was updated within the trial register; 2) We removed the secondary outcome "Ability of the filtering element to inactivate the SARS-Cov-2". The team decided that this outcome would be more appropriately assessed in a controlled laboratory study, and not associated with the clinical trial. Thus, this outcome will be investigated in a secondary study; 3) We decided to include the clinical assessments (Job stress, Quality of life, Musculoskeletal discomfort, Burnout, and Work ability) exclusively as baseline measurements.

ELIGIBILITY:
Inclusion Criteria:

* Full-time employees (defined as direct patient care for more than 24 hours weekly) and work primarily at the study site or co-participants (more than 75% of working hours).
* Professionals working in emergency departments, ICUs, and other hospital settings exposed to SARS-Cov-2.
* Negative clinical and laboratory results for SARS-Cov-2 infection (negative RT-PCR).
* Have previous experience using N95 PFF2 respirators.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* History of high-risk comorbidities, such as high-risk heart disease or respiratory diseases.
* Presence of heterogeneous facial anatomical characteristics such as bulky beard, facial deformities, or facial dimensions incompatible with the respirators.

Ages: 20 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Incidence of laboratory-confirmed COVID-19 | 21 days (Assessments at T1 - day 10, and T2 - day 21)
  Number of professionals infected, confirmed by reverse-transcription polymerase chain reaction (RT-PCR)

SECONDARY OUTCOMES:
Usability and comfort of the respirator | Assessments at T1 (day 10) and T2 (day 21)
  11-point Likert scale ranging from -5 ("extremely unsatisfied"), 0 ("neutral"), to 5 ("completely satisfied")
Adherence to the use of the Respirator | Assessments at T1 (day 10) and T2 (day 21)
  quantified based on the activities and procedures performed by the participants. Adherence will be measured by a self-report recorded in a diary, estimating the percentage of use referring to the total workhours.
Incidence of acute respiratory illness | Change from Pre-Intervention (T0), compared to T1 (day 10), and T2 (day 21)
  Self-reported signs and symptoms of respiratory illness, defined as the presence of at least 1 sign or 2 symptoms (presented to the participants as a list of possible signs and symptoms), and also confirmed by reverse-transcription polymerase chain reaction (RT-PCR).

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo L Carregaro, PhD, Principal Investigator — Universidade de Brasília (FCE/UnB); Suelia S Fleury Rosa, PhD, Study Director — Universidade de Brasília (FGA/UnB); Marcella L Brettas Carneiro, PhD, Study Chair — Universidade de Brasília (FUP/UnB); Henry M Peixoto, PhD, Study Chair — Universidade de Brasília (FM/UnB); Graziella A Joanitti, PhD, Study Chair — Universidade de Brasília (FCE/UnB); Glécia V Silva Luz, PhD, Study Chair — University of Brasilia
Locations (1):
- HRAN (Hospital Regional da Asa Norte), Brasília, Brazil

REFERENCES:
- [Derived] Kubota AMA, Rosa MFF, Baraldi S, Vale JAM, da Silva JDAG, Carneiro MLB, Padula RS, Haddad R, Joanitti GA, da Silva Luz GV, Fook MVL, Zimmermann IR, Rosa SSRF, Peixoto HM, Luiz Carregaro R. Efficacy and feasibility of a novel semi-facial respirator with chitosan nanoparticles on the incidence of SARS-CoV-2 infection in healthcare professionals: randomized controlled trial. BMC Infect Dis. 2024 Sep 27;24(1):1061. doi: 10.1186/s12879-024-09966-x. PMID 39333902